CLINICAL TRIAL: NCT02207517
Title: Convergence Insufficiency Treatment Trial - Attention and Reading Trial (CITT-ART)
Brief Title: Office-based Vision Therapy for Improving Reading and Attention in Children With Convergence Insufficiency
Acronym: CITT-ART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Salus University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Marshall B. Ketchum University (Unknown); Ohio State University (Other); University of Alabama at Birmingham (Other); State University of New York College of Optometry (Other); Akron Children's Hospital (Other); Nova Southeastern University (Other); Bascom Palmer Eye Institute (Other)
Responsible Party: Principal Investigator, Mitchell Scheiman, Dean of Research, Salus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Salus - HMS1310; U10EY022599-01A1 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Convergence Insufficiency
Keywords: convergence insufficiency; vision therapy; reading; attention
MeSH Terms: conditions — Ocular Motility Disorders | interventions — Orthoptics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Office-based verg/accomm therapy (OBVAT) (Experimental): OBVAT requires a participant to undergo a specific vision therapy regimen with 16 weekly, 60-minute in-office treatment sessions. Vision Therapists (O.D., M.D., Orthoptists, or specially-trained technicians) administer the therapy in the office. OBVAT procedures are then supplemented with various home therapy procedures
  Interventions: Procedure: Office-based vergence/accommodative therapy
- Office-based placebo therapy (OBPT) (Placebo Comparator): Office-based Placebo Therapy (OBPT) requires a participant to undergo a specific therapy regimen of 16 weekly, 60 minute, in-office treatment sessions. Vision therapists (optometrists, ophthalmologists, orthoptists, or specially-trained technicians) administer the therapy in the office. OBPT procedures are then supplemented with placebo home therapy procedures.
  The procedures for OBPT are designed with the intent of not providing a beneficial training effect on vergence, accommodation, saccadic accuracy, or visual attention beyond normal activities. However, the procedures are designed to simulate real vision therapy in such a way that it will be difficult for participants and parents to know that they have been assigned to the control group and thus are not receiving bonafide OBVAT
  Interventions: Procedure: Office-based vergence/accommodative therapy

INTERVENTIONS:
Procedure: Office-based vergence/accommodative therapy — The OBVAT program has been divided into 4 phases. Within each phase there are a number of categories such as gross convergence, vergence, and accommodation. The therapy procedures in each category have been arranged sequentially from easiest to most difficult
  Other Names: Vision Therapy; Orthoptics

SUMMARY:
CITT-ART is a multicenter study (8 locations around the United States) of 324 children ages 9 to <14 years with symptomatic convergence insufficiency (CI). The purpose of this study is to see if office-based therapy for convergence insufficiency (CI) improves reading ability and attention. CI is an eye-teaming problem where the eyes would like to drift outward when reading or doing close work. When eyes drift out, double vision can happen. To prevent double vision one must use extra effort to keep the eyes from going out. This extra effort can cause symptoms that can interfere with reading and working comfortably at near. These symptoms often include eyestrain, blurred vision, headaches, double vision, and loss of place when reading or performing tasks at near. In a prior study we found that therapy improves these symptoms. In this study we are looking at whether the therapy improves reading and attention

DETAILED DESCRIPTION:
Following the success of the NEI-funded Convergence Insufficiency Treatment Trials (CITT), the next logical and important research issue is to determine if the successful treatment of symptomatic convergence insufficiency (CI) (i.e., improvement of symptoms and ophthalmic signs) impacts function (reading and attention).

It is well documented that children with symptomatic CI report significantly more symptoms when reading and doing close work (e.g., blurred vision, headaches, double vision, loss of concentration, frequent loss of place, trouble remembering what was read), manifest more academic-impairing behaviors (e.g., difficulty finishing assignments), and score worse on parent ratings of attention compared to children with normal binocular vision. Because reduction of symptoms and adverse academic behaviors are established outcomes of successful treatment of CI, we propose to test the hypothesis that resolution of these symptoms and behaviors leads to improved reading performance and attention. Previous studies have found improvements in reading comprehension reading speed and accuracy after successful treatment of CI. In a recent pilot study, investigators also found significant improvement in reading comprehension and attention after 16 weeks of successful treatment of symptomatic CI with office-based vergence/accommodative therapy; however, there was no control group. To definitively determine whether the successful treatment of symptomatic CI positively impacts reading and attention requires a placebo-controlled randomized clinical trial.

Objective: We propose a multicenter, placebo-controlled, randomized clinical trial (RCT) of 324 children ages 9 to <14 years (Grades 3-8) with symptomatic CI. [we will restrict recruitment to children who do not have significant single word reading deficits.] Participants will be randomized to 16 weeks of treatment with either [a] office-based vergence/accommodative therapy with home reinforcement (OBVAT) or [b] office-based placebo therapy with home reinforcement (OBPT). Outcomes (reading and attention) will be assessed after 16 weeks of treatment. In addition, we will test the long-term effects on outcomes at 1 year after treatment completion. All analyses will test the null hypothesis of no difference in outcomes between the two treatment groups.

Specific Aim 1 - Reading Performance: To compare reading comprehension outcomes for children with symptomatic CI who receive 16 weeks of OBVAT and OBPT treatment. The primary outcome measure of reading performance is the Wechsler Individual Achievement test (WIAT-III) reading comprehension subtest score. In secondary analyses, we will examine the effects of the treatment on word reading, pseudoword decoding, oral reading fluency, and listening comprehension. We also will examine the correlation of changes in CI symptoms and ophthalmic signs with reading outcomes. Analysis of the 1-year follow-up data will be used to determine if any gains in reading performance observed after 16 weeks of treatment are sustained.

Specific Aim 2 - Attention: To investigate the effect of treatment on teacher- and parent-rated measures of attention for children with symptomatic CI who receive 16 weeks of OBVAT and OBPT intervention. The primary outcome measure of attention is the score on the Strengths and Weaknesses of ADHD Symptoms and Normal Behavior Scale (SWAN). In secondary analyses, we will examine the effects of treatment on a second parent-rated attention scale called the SNAP. We also will examine the correlation of changes in CI-symptoms and ophthalmic signs with attention outcomes. Analysis of the 1-year follow-up data will be used to determine if any gains in attention observed after 16 weeks of treatment are maintained.

Scientific and Clinical Impact: The relationship between the treatment of symptomatic CI and its effect on reading and attention in children is unknown. The results of the proposed study will contribute to a better understanding of these relationships and help to resolve controversy surrounding this issue. The results will have important implications for educators, psychologists, eye professionals, and other health care providers who care for children with reading and attention problems and guide hypothesis development for future scientific investigations on evidence-based relationships between visual disorders and other developmental disorders in children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9 to less than 14 years
2. Grades 3 through 8
3. CI Symptom Survey (CISS) score greater or equal to 16
4. Exophoria at near at least 4 prism diopters greater than at far
5. Receded near point of convergence (NPC) of 6 cm or greater break
6. Insufficient positive fusional vergence (PFV) at near (i.e., failing Sheard's or PFV less than or equal to 15 BO break)
7. Best-corrected distance visual acuity of 20/25 or better in each eye
8. Random dot stereopsis appreciation of 500 seconds of arc or better
9. Wearing appropriate refractive correction (spectacles or contact lenses) for at least 2 weeks prior to final determination of eligibility for any of the following uncorrected refractive errors (based on cycloplegic refraction within prior 12 months)

   * Myopia greater than -0.75D spherical equivalent (SE) in either eye
   * Hyperopia greater than +2.00D SE in either eye
   * SE anisometropia greater than 0.75D
   * Astigmatism greater than 1.00D in either eye

   Correction for patients meeting above refractive error criteria must meet the following guidelines:
   * SE anisometropia must be within 0. 75D of the full anisometropic correction
   * Astigmatism must be within 0.75D of full correction; axis must be within 6◦ if astigmatism greater than or equal to 1.00D
   * For hyperopia, the sphere can be reduced by up to 1.50 D provided reduction is symmetrical
   * For myopia, the SE must be within 0.75D of the full myopic correction
10. No use of BI prism or plus add at near for 2 weeks prior to study and for duration of study
11. English is primary language spoken at home or child proficient in English as determined by the school
12. Parent does not expect child to start any new ADHD medicine or change the dose of any currently taken ADHD medicine while child is being treated in the study
13. Parental permission to contact the child's teacher(s) for study purposes
14. Parent and child understand protocol and are willing to accept randomization

Exclusion Criteria:

1. Constant strabismus at distance or near
2. Esophoria of greater than or equal to 2∆ at distance
3. Vertical heterophoria greater than or equal to 2∆ at distance or near
4. greater than or equal to 2 line interocular difference in best-corrected distance visual acuity
5. Monocular near point of accommodation greater than 20 cm (accommodative amplitude less than 5D) in right eye
6. Manifest or latent nystagmus
7. Word Reading subtest score less than 80 on the Wide Range Achievement Test (WRAT-4)
8. Kaufman Brief Intelligence Test (KBIT-2) Matrices subtest score less than 70
9. History of prior strabismus, intraocular, or refractive surgery
10. CI previously treated with any form of office-based vergence/accommodative therapy or home-based vergence therapy (e.g., computerized vergence therapy)
11. CI associated with head trauma or known disease of the brain
12. Diseases known to affect accommodation, vergence, or ocular motility
13. Inability to comprehend and/or perform any study-related test or therapy procedure
14. Speech-language disorder (e.g., stuttering) that would interfere with interpretation of digital recordings of reading tests
15. Significant hearing loss
16. Household member enrolled in present CITT-ART, treated currently, or treated within the past 6 months with any form of office-based vergence/accommodative therapy or home-based vergence therapy (e.g., computerized vergence therapy)
17. Parent or other household member is an eye care professional, ophthalmic technician, ophthalmology or optometry resident, or optometry student

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
The change in the Wechsler Individual Achievement Test-III (WIAT-III) reading comprehension score as measured after the completion of 16 weeks of assigned treatment (OBVAT or OBPT). | After 16 weeks of treatment
  This test requires the examinee to respond to multiple-choice questions after having read passages independently.

SECONDARY OUTCOMES:
The change in the Strengths and Weaknesses of ADHD Symptoms and Normal Behavior Scale (SWAN) | After 16 weeks of treatment
  The SWAN is a behavior rating scale that has been used for many years as an assessment tool for ADHD.
Gates-McGintie 4 | After 16 weeks of treatment
  The child must respond to multiple-choice questions after having read passages independently
d2 Test of Attention | After 16 weeks of treatment
  The d2 is a timed test of selective and sustained attention.The test measures processing speed, rule compliance, and quality of performance in response to the discrimination of similar stimuli, thereby allowing for an estimation of individual attention and concentration performance
Academic Behavior Survey (ABS) | After 16 weeks of treatment
  The ABS is a 6-item survey designed to measure the frequency of adverse academic behaviors and parental worry about academic performance.
Curriculum Based Measurement (CBM) | After 16 weeks of treatment
  Curriculum Based Measurement is commonly used by educators to assess short-term progress in reading, skills as the child proceeds through the academic year The primary advantage of the CBM measure is the ability to track rate of improvement by initial reading level and by time of year. The addition of the CBM measure will assess reading at each outcome visit and allow us to track changes in a similar manner to attention and CI where we have measures at each outcome visit. In addition, CBM will provide an additional outcome measure for reading using a method that is commonly employed by school districts to monitor reading progress and will help to communicate the clinical significance of our results.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, OD, Study Chair — Salus University; Lynn MItchell, MAS, Principal Investigator — Ohio State University
Locations (8):
- United States (8):
  - University of Alabama, Birmingham College of Optometry, Birmingham, Alabama
  - Southern California College of Optometry Marshall B. Ketchum University, Fullerton, California
  - NOVA Southeastern University College of Optometry, Fort Lauderdale, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - State University of Optometry College of Optometry, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Ohio State University College of Optometry, Columbus, Ohio
  - Pennsylvania College of Optometry at Salus University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] CITT-ART Investigator Group. Effect of Vergence/Accommodative Therapy on Attention in Children with Convergence Insufficiency: A Randomized Clinical Trial. Optom Vis Sci. 2021 Mar 1;98(3):222-233. doi: 10.1097/OPX.0000000000001659. PMID 33771952
- [Derived] Scheiman M, Kulp MT, Cotter SA, Lawrenson JG, Wang L, Li T. Interventions for convergence insufficiency: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 2;12(12):CD006768. doi: 10.1002/14651858.CD006768.pub3. PMID 33263359
- [Derived] CITT-ART Investigator Group. Effect of Vergence/Accommodative Therapy on Reading in Children with Convergence Insufficiency: A Randomized Clinical Trial. Optom Vis Sci. 2019 Nov;96(11):836-849. doi: 10.1097/OPX.0000000000001442. PMID 31651592